CLINICAL TRIAL: NCT05718206
Title: Research on Diagnosis and Prognosis of Myocardial Ischemia Level in Xiangya Hospital Using Magnetocardiography -- Miracle MCG
Brief Title: Research on Diagnosis and Prognosis of Myocardial Ischemia Level Using Magnetocardiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202209584
Record Dates: First submitted 2022-12-25; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Stable Ischemic Heart Disease; Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia | interventions — Magnetocardiography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronary stenosis (Experimental)
  Interventions: Device: Magnetocardiography
- Control (Other)
  Interventions: Device: Magnetocardiography

INTERVENTIONS:
Device: Magnetocardiography — Both arms underwent magnetocardiogram examination, and three experts interpreted magnetocardiogram results independently.

SUMMARY:
Magnetocardiography (MCG) is a non-invasive and accurate method of detecting myocardial ischemia. However, the previous MCG is limited in clinical practice due to its high working conditions and limited sensitivity. The next-generation MCG based on optical pumped magnetometer (OPM) has the advantages of high sensitivity, high reliability, high usability and low cost, which makes it suitable for most medical scenarios. Thus, this prospective single-center study aimed to use OPM MCG to explore its diagnostic efficacy and predictive value for myocardial ischemia. Participants who will receive coronary angiography examinations will be enrolled in this study. Participants enrolled in the study will also have a 1, 3, 6, 12, 24, 36, and 48-month follow-up for analysis of adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Those who are suspected of coronary heart disease and scheduled to undergo coronary angiography;
3. Sign the informed consent.

Exclusion Criteria:

1. Complex arrhythmia, including frequent premature atrial beats, premature ventricular beats, atrial fibrillation, atrial flutter, and complete bundle branch block;
2. Severe hypertension (> 180/110 mmHg);
3. Congenital heart diseases, valvular heart diseases, or implantation of pacemakers or drug pumps.
4. Severe thoracic or pulmonary diseases, thoracic malformation, or history of thoracic surgery;
5. Pregnant or breastfeeding women;
6. Claustrophobia, or those who can't lie still for 2 minutes in a confined space;
7. Allergy to contrast agent;
8. Renal impairment: serum creatinine > 2,0 mg/dl (176.8 μmol/L) or those who are receiving hemodialysis;
9. Other diseases, including malignant tumors, organ transplantation, and candidates for organ transplantation;
10. History of alcohol or drug abuse (cocaine, heroin, etc.);
11. Participating in clinical studies of other drugs or devices without reaching the time limit for the primary endpoint;
12. Those who aren't suitable for inclusion due to other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-08-14 (Estimated); Study Completion 2025-08-14 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of diagnosis of myocardial infarction level | up to 6 months
  The myocardial ischemic level is measured by MCG and coronary angiography examination. The result of the coronary angiography examination is independently judged by three experienced clinicians. And calculate the sensitivity to evaluate the diagnosis of myocardial infarction level validity.
Specificity of diagnosis of myocardial infarction level | up to 6 months
  The myocardial ischemic level is measured by MCG and coronary angiography examination. The result of the coronary angiography examination is independently judged by three experienced clinicians. And calculate the specificity to evaluate the diagnosis of myocardial infarction level validity.
Consistency of diagnosis of myocardial infarction level | up to 6 months
  The myocardial ischemic level is measured by MCG and coronary angiography examination. The result of the coronary angiography examination is independently judged by three experienced clinicians. Calculate the consistency to evaluate the diagnosis of myocardial infarction level reliability.
Kappa statistics of diagnosis of myocardial infarction level | up to 6 months
  The myocardial ischemic level is measured by MCG and coronary angiography examination. The result of the coronary angiography examination is independently judged by three experienced clinicians. Calculate the Kappa statistics to evaluate the diagnosis of myocardial infarction level reliability.

SECONDARY OUTCOMES:
Incidence of major adverse cardiovascular events | through study completion, an avarage of 2 years
  Participants are followed up by telephone at 1, 3, 6, 12, 24, 36, 48, and 60 months after recruitment and ask whether major adverse cardiac events (MACE) have happened. MACE will be defined as acute myocardial infarction, coronary revascularization, stroke, and all-cause death. According to incidence of MACE, draw the Kaplan-Meier curve and establish Cox regression model.Establish a risk-predicted model of MCG for detecting myocardial infarction